CLINICAL TRIAL: NCT00496808
Title: Neoadjuvant Herceptin for Ductal Carcinoma In Situ of the Breast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0701
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2012-05-18 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Ductal Carcinoma In Situ
Keywords: Ductal Carcinoma In Situ; Breast Cancer; Herceptin; Trastuzumab; DCIS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Herceptin (Experimental): 8 mg/kg intravenously (IV) Over 90 Minutes
  Interventions: Drug: Herceptin (Trastuzumab)

INTERVENTIONS:
Drug: Herceptin (Trastuzumab) — 8 mg/kg IV Over 90 Minutes
  Other Names: Trastuzumab

SUMMARY:
Primary Objectives:

* To determine the effect of a single dose of Herceptin (trastuzumab) on the proliferation rate of Her-2/neu over-expressing ductal carcinoma in situ (DCIS)
* To evaluate the effect of a single dose of Herceptin on the apoptotic index of Her-2/neu over-expressing DCIS

DETAILED DESCRIPTION:
Herceptin (Trastuzumab) stops or slows the growth of certain breast cancer cells by blocking the chemical signals they need to grow.

As part of your standard care for DCIS, you will have a complete routine physical exam, a mammogram of both breasts, and blood (about 2 tablespoons) will be drawn for routine tests. Some of your leftover breast biopsy tissue will be tested for Her-2/neu expression. Blood will be drawn (about 2-6 teaspoons) to check if your bone marrow (red blood cells), kidney, and liver are functioning well enough to have this treatment. Women who are able to have children must have a negative blood pregnancy test before starting treatment.

If you are eligible to take part in this study, you will receive one dose of trastuzumab at least 2 weeks before your surgery. The dose of trastuzumab will be given intravenously (through a needle in a vein in your arm) as a steady infusion over 90 minutes, on an outpatient basis. You will be checked during the infusion and for 1 hour after it is completed.

You will have routine surgery for DCIS (either segmental mastectomy, mastectomy with or without reconstruction, and possible sentinel lymph node biopsy) approximately 14 to 28 days after being given Herceptin. If a segmental mastectomy was performed as part of our standard practice you will be evaluated by a radiation oncologist following surgery. After your surgery, patients will also be evaluated by a breast medical oncologist to determine if any additional standard therapy is needed.

Tissue that is left over from the original breast biopsy and surgery will be tested for various biomarkers (substances which indicate the severity or spread of cancer), cancer growth rate, and apoptotic index (cell death rate).

This is an investigational study. The FDA has approved trastuzumab for the treatment of breast cancer. Up to 71 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with histologic confirmation of DCIS (TisN0M0) that is Her-2/neu 3+ positive by immunohistochemistry (IHC) and/or positive for Her-2 gene amplification by fluorescence in situ hybridization (FISH) will be eligible for the study.
2. Patients must sign informed consent indicating that they are aware of the investigational nature of the study, in keeping with institutional policy.
3. Those patients with history of other contralateral non-invasive and invasive breast and non-breast malignancies are eligible to participate unless they have previously received a doxorubicin dose of more than 400 mg/m2.
4. All patients should have adequate bone marrow function, as defined by peripheral granulocyte count of > 1,500/mm3, and platelet count > 100,000 mm3. Patients must have adequate liver function, with bilirubin within normal laboratory values. In addition, patients should have adequate renal function, defined as serum creatinine < 2.0 mg/dl.
5. Patients with intact primary tumors will be eligible for this study. Patients who have had their diagnostic biopsy at an outside facility but still have measurable disease on presentation will be eligible.
6. Patients with history of cardiac arrhythmia will be eligible for study after being seen by cardiology and deemed good candidates for participation.
7. Women of child bearing potential must have a negative urine or serum pregnancy test.

Exclusion Criteria:

1. Patients with a current known invasive breast cancer are not eligible for this study.
2. All patients who are Her-2/neu negative will be ineligible for the study.
3. Patients with history of congestive heart failure will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Kuerer, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2005 - November 2010. All recruitment was at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Herceptin
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Herceptin
Number analyzed (Participants) | 69
Age, Continuous [Median (Full Range); unit: years] | 53 [31 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Proliferation as Measured by Ki-67
Description: Percent Change in Proliferation as measured by Ki-67 (% nuclei stained). Comparison of proliferation rates of Her-2/neu overexpressing cells before and after treatment with Herceptin per Participant where absolute change defined as difference of increase/decrease. Proliferation rate evaluated by immunohistochemistry using paraffin-embedded sections and monoclonal antibody for ki-67.
Time Frame: Before and after single dose of Herceptin approximately 21 days before surgery for ductal carcinoma in situ (DCIS), up to 4 weeks
Reporting Status: Not Posted

2. Primary Outcome: Number of Participants Achieving Documented Change in Proliferation
Description: Proliferation rate and apoptotic index measured on core biopsy specimen and resection specimen from each participants. To compare Antibody-Dependent Cell-Mediated Cytotoxicity (ADCC) and CD4+ T-cell response in each participant observed at pre- and post-treatment times, paired analysis was performed using Student's t-test. Nonparametric Wilcoxon rank sum test was used to compare data between groups.
Time Frame: Before and after single dose of Herceptin approximately 21 days before DCIS surgery, up to 4 weeks
Population: Twelve evaluable patients were required to characterize the change in proliferation rate after treatment with a single dose of Herceptin (trastuzumab). Those participants who completed Herceptin administration, surgery, and post surgery bio-markers testing were evaluable.
Measure: Number; unit: Participants
Arm/Group | Herceptin
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Mean Percent of Ki-67
Description: Mean percent of Ki-67 (% nuclei stained) at immunohistochemical staining performed for biomarkers. Tissue sections from diagnostic core biopsy tissue that contains DCIS before treatment and from corresponding tissues that contain DCIS from the surgical resection obtained after a single dose of Herceptin.
Time Frame: Before and after single dose of Herceptin approximately 21 days before DCIS surgery, up to 4 weeks
Population: Analysis was per protocol. Twelve evaluable patients were required to characterize the change in proliferation rate after treatment with a single dose of Herceptin (trastuzumab). Those participants who completed Herceptin administration, surgery, and post surgery bio-markers testing were evaluable.
Measure: Mean (Standard Deviation); unit: Percentage of Ki-67
Arm/Group | Herceptin
Number analyzed (Participants) | 12
Percentage of Ki-67 | 44.29 (3.42)

ADVERSE EVENTS:
Time Frame: 3 years and 2 months
Arm/Group | Herceptin
Serious Adverse Events (participants affected / at risk) | 3/69
Other Adverse Events (participants affected / at risk) | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Herceptin (N=69)
Infusion reaction (General disorders) | 2 (2) — Grade I or II consisting of chills or chills and fever resolve with diphenhydramine and acetaminophen or hydrocortisone and meperidine respectively
Neuropathy: Sensory (Nervous system disorders) | 1 (1) — Parasthesia to right side of face and lip with tingling sensation not interfering with function

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes